CLINICAL TRIAL: NCT03295981
Title: Local Bisphosphonate Effect on Recurrence Rate in Extremity Giant Cell Tumor of Bone: A Prospective Randomized Controlled Trial
Brief Title: Local Bisphosphonate Effect on Recurrence Rate in Extremity Giant Cell Tumor of Bone
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: St. Louis University (Other)
Collaborators: Orthopedic Research and Education Foundation (Other); Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other); University of Iowa (Other); Johns Hopkins University (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); The Cleveland Clinic (Other); Wake Forest University (Other); University of Kansas (Other); Indiana University (Other); University of Oklahoma (Other); Beth Israel Deaconess Medical Center (Other); Boston Children's Hospital (Other); American Academy of Orthopaedic Surgeons (Other); Massachusetts General Hospital (Other); All India Institute of Medical Sciences (Other); University of Washington (Other); University of California (Other)
Responsible Party: Principal Investigator, David Greenberg, MD;; Associate Professor, Professor Orthopaedic Surgery Saint Louis University, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 28229
Record Dates: First submitted 2017-09-18; First posted 2017-09-28 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Giant Cell Tumor of Bone
MeSH Terms: conditions — Giant Cell Tumor of Bone | interventions — Zoledronic Acid

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control group (No Intervention): The surgical procedure for all patients will include extensive curettage of the lesion to remove macroscopic tumor, high-speed burring of the residual cavity, adjuvant treatment to the residual cavity, followed by packing of the cavity with either polymethylmethacrylate (PMMA) bone cement (Simplex P; Stryker, Mahwah, New Jersey) alone or bone cement with subchondral allograft bone graft. The choice of cavity reconstruction will be at the discretion of the treating surgeon. Traditional local adjuvants (argon beam coagulation, phenol, ethanol, or cryotherapy) will be used depending on surgeon preference. In addition to the above standard treatment, the patients will be randomized into one of two study arms. In Arm 1, the control group, no additional local therapy will be utilized.
- Bisphosphonate group (Experimental): In Arm 2, the bisphosphonate group, 4 mg of zoledronic acid (Zometa) will be added to each bag of bone cement.
  Interventions: Drug: Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic Acid — 4 mg of zoledronic acid (Zometa) will be added to each bag of bone cement
  Other Names: zoledronate
  Arms: Bisphosphonate group

SUMMARY:
The purpose of the clinical study is to investigate whether the local delivery of bisphosphonate as a surgical adjuvant can decrease the chance of a giant cell tumor of bone coming back to the same location. The hypothesis is that the local administration of bisphosphonate will decrease the rate of the tumor returning compared to traditional aggressive surgical removal of the tumor.

DETAILED DESCRIPTION:
The purpose of the clinical study is to investigate whether the local delivery of bisphosphonate (BP-loaded PMMA bone cement) as a surgical adjuvant can decrease the local recurrence rate of giant cell tumor (GCT) of bone. The investigators will evaluate whether bisphosphonate as a surgical adjuvant improves secondary outcomes, such as pain, function, fever, or wound complications. The hypothesis is that the local administration of bisphosphonate will decrease the recurrence rate of GCT compared to traditional aggressive intralesional curettage.

ELIGIBILITY:
Inclusion Criteria:

* Primary benign GCT of bone
* Lesion located in an extremity
* Lesion amenable to reconstruction (intralesional curettage) defined as having at least one intact column of bone after removal
* No previous systemic bisphosphonate or denosumab therapy

Exclusion Criteria:

* Recurrent GCT of bone
* Non-extremity location
* Lesion too extensive for intralesional treatment, either due to bone loss, joint invasion, or large soft tissue component
* Children and pregnancy
* Previous systemic bisphosphonate or denosumab therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-05-03 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
The endpoint for patient participation will be local recurrence | Followed for 2 years postoperatively for study end points
  Local recurrence of giant cell tumor of bone

SECONDARY OUTCOMES:
MSTS Score | Followed for 2 years postoperatively for study end points
  The Musculoskeletal Tumor Society (MSTS) scoring system is a validated and well-accepted functional scoring system used in orthopaedic oncology research
Surgical site infection | Follow-ups will consist of clinical visits. The clinical visits will be at 2 weeks postoperatively, 6 weeks postoperatively, and then every three months for the first two years after surgery.
  The surgical site will be assessed for a surgical site infection (SSI) as defined by CDC guidelines after surgery and during scheduled follow-up as outlined in time frame below.
Wound healing | Follow-ups will consist of clinical visits. The clinical visits will be at 2 weeks postoperatively, 6 weeks postoperatively, and then every three months for the first two years after surgery.
  The surgical site will be assessed after surgery and during scheduled follow-up as outlined in time frame below for wound healing issues/concerns.
Potential bisphosphonate complications related to systemic administration | Followed for 2 years postoperatively for study end points
  Patients will be followed for atypical femur fractures and avascular necrosis (AVN) of jaw

CONTACTS AND LOCATIONS:
Locations (16):
- United States (14):
  - University of California - Los Angeles, Los Angeles, California
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas, Overland Park, Kansas
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Saint Louis University, St Louis, Missouri
  - Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - University of Washington, Seattle, Washington
- McGill University Health Centre, Montreal, Quebec, Canada
- All India Institute of Medical Science, New Delhi, India

IPD SHARING:
Plan to Share IPD: No